CLINICAL TRIAL: NCT03849924
Title: Promoting and Protecting Subjective Well-Being Using Self-Affirmation
Brief Title: Enhancing One's Sense of Self Using Self-Affirmation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Charlotte Entwistle, Research Assistant, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NHS001384
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Mental Health Wellness 1; Anxiety; Self Esteem
Keywords: well-being; randomised controlled trial; intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to an intervention group, intervention 'booster' group (receive the intervention twice) or a control group via a web-based randomiser.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The questionnaire administrator/investigator and participants are blind to the condition, as participants are not informed of the questionnaires being different from one another, and participants should return their questionnaires in sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-affirmation (Experimental): Participants assigned to the self-affirmation intervention condition will undergo a self-affirmation intervention in the form of a questionnaire at time point one (one week after the intervention). This is a brief intervention that involves forming self-affirming implementation intentions. Implementation intentions are formulated plans that encourage one to link critical situations with appropriate behavioural responses. In this study participants are encouraged to write out the stem and their response to the stem from the four options.
  Interventions: Behavioral: Self-affirmation
- Self-affirmation 'booster' (Experimental): Participants assigned to this condition will undergo the self-affirmation intervention described above twice, in comparison to just once, in the form of a questionnaire at time points one (one week after the intervention) and two (two weeks after the intervention).
  Interventions: Behavioral: Self-affirmation
- Control (No Intervention): Participants assigned to the control condition will not undergo a self-affirmation intervention. Instead they will still complete the same questionnaire as participants in the intervention conditions but without the self-affirmation intervention included (normally included on the last page of the questionnaire).

INTERVENTIONS:
Behavioral: Self-affirmation — Self-affirmation implementation intentions in the form of a questionnaire.
  Arms: Self-affirmation; Self-affirmation 'booster'

SUMMARY:
This study evaluates whether a brief psychological intervention, known as a self-affirmation intervention which works by allowing one to recognise their own value, can improve well-being. This study also evaluates whether more of these interventions will lead to greater increases in well-being, and also measures self-esteem and anxiety to examine their potential involvement in the self-affirmation process. Participants are randomly assigned to either a self-affirmation intervention group, a 'booster' self-affirmation group whereby they receive the intervention twice, or a control group (no intervention). Participant's well-being, self-esteem and anxiety are assessed at baseline (before the intervention), 1 week, and 2 weeks after the intervention. It is hypothesised that those who undergo self-affirmation will have more improved levels of well-being than those who do not; those who undergo the self-affirmation twice will have the most improved levels of well-being. It is also hypothesised that self-esteem and state anxiety will be involved in the self-affirmation process and potentially mediate the effects of self-affirmation on well-being.

DETAILED DESCRIPTION:
Subjective well-being, refers to an appraisal of one's own life as a whole. Subjective well-being is regularly being used by governments as a measure of observing social progress, informing new policy and promoting behaviour change, in comparison to more objective measures of social progress such as gross domestic product. A key aim of government policies is therefore to find the most efficient, cost-effective ways to improve people's subjective well-being, to determine the most efficient ways of improving quality of life. There are currently a number of ways in which the government is attempting to address this, with programs in place that are designed to improve people's well-being, such as Altogether Better (Yorkshire and Humber Strategic Health Authority) and Target Well-being (Federation of Groundwork Trust), as well as NHS programmes and free well-being courses. However, these programmes were not always found to be effective in improving people's well-being, particularly when the programmes involved health awareness activities. This limited effectiveness of programmes involving health awareness activities makes them unlikely to be cost-effective as a well-being intervention. This suggests the importance of developing an effective intervention to improve people's well-being, that could also be used within government/NHS well-being programs, to enhance the effectiveness of said programs in improving well-being to make them more cost-effective, particularly in those promoting health awareness.

Self-affirmation theory provides an approach to improve subjective well-being by overcoming feelings of threat to the self. A threat to one's sense of self could undermine one's subjective well-being. Self-affirmation theory states that people strive to maintain a positive, moral and adaptive self-image, and that threats to the self (e.g., a smoker being told that smoking is bad for them), motivates them to defend their global sense of self (e.g., by convincing themselves that the information is flawed). According to self-affirmation theory, people's sense of self can also be protected by bolstering self-image in a domain that is not under direct threat. For example, if one feels that their sense of self is threatened in a certain domain (e.g., by anti-smoking messages), then one can bolster self-image by compensating in another domain (e.g., by doing charity work). There is a large amount of evidence to support this theory, mostly from studies in which self-affirmation manipulations (i.e. by reminding people of their 'core values') have been found to be effective in overcoming threats to the self and promoting receptiveness to health-risk communications.

The effectiveness of self-affirmation in overcoming threats to the self is not specific to health-risk communications as research has found self-affirmation also to be effective in overcoming threats to the self that occur within other domains, such as self-esteem, anxiety and well-being, suggesting that they could be employed to protect subjective well-being across populations at a low cost. There are limitations associated with research in this area however, as there have only been very few studies that have looked at the effects of self-affirmation on well-being and their samples are often limited and lack generalisability. Also, no research to date has measured whether more self-affirmation interventions would produce greater effects. This is of importance as research has regularly demonstrated evidence of dose dependant relationships between a psychological intervention and its subsequent effects, with a greater number of psychological interventions being associated with greater effects. It would also be beneficial if research were to be conducted to determine the effects of self-affirmation in a sample of people who are already undergoing a well-being intervention (e.g., a government programme or NHS course), to see whether self-affirmation can enhance the effectiveness of the intervention in improving well-being, as this has not yet been explored and could help to make the intervention more cost-effective. Therefore, the present study aims to confirm this positive effect of self-affirmation on subjective well-being in a sample that consists of a wider range of backgrounds and demographics that are already undergoing a well-being intervention.

In addition to this, there has been research that has looked at examining mediators of the self-affirmation process, however the mechanisms for explaining the effects of self-affirmation are not yet clearly understood. Some research has found evidence of self-esteem acting as a mediator in the self-affirmation process. However, more research needs to be conducted to confirm these findings as they have been inconsistent, with some research showing no evidence of self-esteem acting as a mediator. Furthermore, other research has found that self-affirmation led to reductions in state anxiety. This suggests state anxiety may be acting as a mediator in the self-affirmation process, as undergoing self-affirmation resulted in changes in state anxiety, with the self-affirming effects possibly being occurring due to reductions in state anxiety. As there has been no research that has addressed this possibility of state anxiety acting as a mediator in the self-affirmation process, research should be conducted on this as this as this would allow greater understanding of the mechanisms involved.

Accordingly, the present study will test the ability of self-affirmation to promote and/or protect subjective well-being by comparing differences in subjective well-being in those that undergo self-affirmation interventions with those that do not. The study will also compare the difference between the effects of one self-affirmation intervention with that of two self-affirmation interventions (i.e. the 'booster' condition), to determine whether there is a dose-dependent relationship of the effects of self-affirmation. The present study will also measure the effects of self-affirmation on self-esteem and state anxiety to test the possibility of mediators of the self-affirmation process. Participants will be recruited from an NHS college which runs free courses that are designed to help people improve their health and/or well-being. It is likely that those who attend this college may feel threatened by the courses, such as feeling threatened by opening-up and talking through issues during the courses, which would lead to defensive processing and undermine the effectiveness of the courses in their aim of improving people's well-being. Self-affirmation could help to overcome these feelings of threat by reducing defensive processing, which could then enhance the effectiveness of the courses in helping people improve their well-being. This is a particularly important population to recruit from as the courses ran by the college often promote health awareness, which research has identified as being less effective in improving well-being. Self-affirmation interventions could therefore help to improve the cost-effectiveness of the courses.

The present study has three aims; the first aim is to confirm previous findings that brief self-affirmation interventions can enhance and protect subjective well-being, in a sample of people already undergoing a well-being intervention, to see whether self-affirmation can enhance the effectiveness of the intervention. The second aim is to examine the possibility of mediators involved in producing the effects of self-affirmation, namely state anxiety, self-esteem and self-esteem domains, to increase understanding of the mechanisms involved in the self-affirmation process. State anxiety and self-esteem have been decided upon due to the inconsistent findings surrounding self-esteem acting as a mediator of self-affirmation and the lack of research on state anxiety acting as a mediator of self-affirmation. The third aim is to measure whether this effect of self-affirmation on subjective well-being is greater in those that undergo a greater number of self-affirmation interventions, as to whether or not there is a dose-dependent relationship between self-affirmation and its' effect on subjective well-being. This could then be used in practice to further enhance the positive effects of self-affirmation, by providing more self-affirming interventions for example. It is hypothesised that there will be higher levels of subjective well-being, after controlling for baseline scores, in those that receive a self-affirmation intervention compared to those that do not. Also, this effect will be greater, with more improved levels of subjective well-being, in those that receive the self-affirmation intervention twice compared to those that only receive it once. This is hypothesised due to findings from research in other domains of more psychological interventions producing greater effects; known as a dose-dependent relationship. It is also hypothesised self-esteem and state anxiety will act as mediators in the self-affirmation process, based on previous findings of relationships between them and self-affirmation.

Participants- Based on the medium effect size of f = 0.25 for a within/between-participants MANOVA of three levels and three dependent variables, G-power software was used to conduct a power analysis to calculate the required sample size. A medium effect size was used for this analysis as there has been little previous research on self-affirmation in which there were three levels of the between participants factor and three dependant variables. As the analysis required an F-test with a between-factors MANOVA with three levels, also assuming an error probability of 0.05 and a statistical power of 0.80, it presented a required sample size estimated to be N = 81.

Accordingly, this study aimed to recruit a total of 100 participants to allow for attrition. This was calculated based on findings of a median retention rate (participants that had completed baseline and follow-up) of 89% from 151 longitudinal randomised control trials (RCT). However, these RCT's were clinical trials in which participants were often offered incentives for participating, with follow-up regularly being retrieved from medical files, as 84% of all trials were conducted in a hospital or general practice (GP) setting. Therefore, as the participants in the present study were not offered any incentives for participation and the study is not being carried out in a hospital setting, there are likely to be higher attrition rates when compared to those calculated based on previous RCT's. To account for this likelihood of higher attrition rates, the initial participant recruitment aim of 90 participants was rounded up to 100 participants.

Participants are to be recruited via opportunity sampling from an NHS college, in the North-West area of England, which runs a variety of free courses lasting from 2-8 weeks. These courses aim to enhance people's health and well-being. Examples of the courses run by the college include courses on improving sense of control, recovery from depression and anger management. Participants will be recruited from this college as it is likely that those who attend these college courses may feel threatened by the nature of the courses, by having to talk through personal issues during the courses for example, which may then inhibit the effectiveness of the courses in improving well-being. The present study therefore recruited people from this college in order to see whether self-affirmation could help people to overcome feelings of threat generated by the courses, and so enhance the effectiveness of the courses in improving well-being; increasing the cost-effectiveness of the courses. Participants will not be offered any incentives for participating in the study.

Proposed Analysis- To measure the effectiveness of the randomisation procedure a MANOVA, using SPSS, will be conducted. The independent variable will be condition with 3 levels: 'standard' self-affirmation, 'booster' self-affirmation and a control. The dependant variables will be age, gender and baseline measures of subjective well-being, self-esteem and state anxiety. If the multivariate and univariate tests are non-significant then this will demonstrate that the participants were successfully randomised to the conditions.

To measure the effects of self-affirmation on subjective well-being a mixed 3 x 3 ANOVA, using SPSS, will be conducted. The between-participants factor will be condition with 3 levels ('standard' self-affirmation vs 'booster' self-affirmation vs control), and the within participants factor will be time with 3 levels (baseline assessment vs 'booster' assessment vs follow-up assessment). The dependent variable will be subjective well-being. An ANCOVA will be conducted to explore any significant interactions. For the ANCOVA, the between-participants factor will be condition, the dependent variable will be follow-up scores and the covariate will be baseline scores. Mediator analysis will also be conducted to examine whether self-esteem and state anxiety act as mediators in the self-affirmation process. This will be done using R software via the 'mediation' package.

Ethical Considerations- Ethical approval has been granted via HRA and REC ethics. Participants will be informed that by completing and handing in the questionnaire they are consenting to participate in the study. Participants will be informed that they do not have to participate in the study if they do not want to and they can choose to withdraw from the study, and withdraw their data, at any time. Participants will also be informed that their data will remain anonymous and confidential as participants' names, and any other identifiable information, will not be required.

Due to the follow-up nature of the study, the participants' baseline and follow-up questionnaires will need to be matched. In order to match the participants' two questionnaires, whilst keeping their data anonymous and confidential, they will be asked to create an identifiable code and state this on both questionnaires. Data storage will comply with the requirements of the Data Collection Act 1998. All manual data (i.e. participant questionnaires) will be immediately transferred onto a protected university computer, by copying the data onto an Excel spreadsheet once the data has been collected. The manual data will be shredded immediately after it has been transferred onto the protected university computer. All data will be stored on the protected university computer under password protected folders and removed once the 5-year data storage period ends, via deleting the files and removing them from the recycling bin, only the chief and principal investigators will have access to the protected university computer. Study data and material may be looked at by individuals from the University of Manchester, from regulatory authorities or from the NHS Trust, for monitoring and auditing purposes.

Although participants will originally be informed that the questionnaires are assessing personal and social beliefs, participants will be verbally debriefed on the true nature of the study by the principal investigator, after the follow-up questionnaires have been completed. Not informing participants of the true nature of the study, that it will involve using self-affirmation, is necessary as research has found that awareness of the self-affirmation process may diminish its impact. Participants' demographic variables will also be assessed (e.g., age, gender, income), which some may find intrusive. However, participants will be advised that they do not have to provide this information if they do not wish to and instead they can leave this blank. Appropriate contact details from the University of Manchester will be provided to participants to allow them to contact someone if they have any issues surrounding the research, during or after the study.

ELIGIBILITY:
Inclusion Criteria:

* Anyone that attends the NHS college designed to improve health and well-being that is willing to participate in the study

Exclusion Criteria:

* Any cognitive/psychological deficits that would affect the individual's capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline subjective well-being at 2-weeks follow up | Through study completion, up to 2 weeks
  This questionnaire assesses the three main components of subjective well-being, using the four items advised by the UK Office for National Statistics. These subjective well-being components include evaluation ("Overall, how satisfied are you with your life nowadays?"), experience ("Overall, how happy did you feel yesterday?" and "Overall, how anxious did you feel yesterday?") and eudemonic ("Overall, to what extend do you feel the things you do in your life are worthwhile?"). Participants were asked to respond to questionnaire items on 11-point Likert-type scales from 'not at all' (0) to 'completely' (10).

SECONDARY OUTCOMES:
Change from baseline self-esteem at 2-weeks follow up | Through study completion, up to 2 weeks
  Robins et al.'s (2001) scale- This scale only consists of one item, namely "I have high self-esteem".
Change from baseline self-esteem domains at 2-weeks follow up | Through study completion, up to 2 weeks
  Another self-esteem measure that was used in the study is Geller et al.'s, (1997) shape and weight-based self-esteem scale. This was used to determine the domains of which participants derive their self-esteem from. Participants were presented with a list of 8 items, from 8 domains, of which they may derive their self-esteem from. They were then asked to identify which domains are important to them and then rank these in terms of their personal importance.
Change from baseline state anxiety at 2-weeks follow up | Through study completion, up to 2 weeks
  Marteau and Bekker's (1992) short version of the state scale of the Spielberger State-Trait Anxiety Inventory (1979) was used to measure state anxiety. It consists of six items on 4-point Likert-type scales ranging from 'not at all' (1) to 'very much' (4). The six items used in the inventory are "I feel calm", "I am tense", "I feel upset", "I am relaxed", "I feel content" and "I am worried".

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte S Entwistle, MRes, Principal Investigator — University of Manchester
Locations (1):
- Pennine Care NHS Foundation Trust- The Health and Well-being College, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT03849924/Prot_SAP_000.pdf